CLINICAL TRIAL: NCT02790424
Title: Adjustment Exploratory Protocols (MagnetoEncephaloGraphy Study : MEG, ElectroEncephaloGram : EEG, Magnetic Resonance Imaging : MRI, Functional MRI : MRIf, Motor Platform) and Functional Evaluation of New Non Invasive Devices (REX BIONICS Exoskeleton) in Patient Volunteers
Brief Title: Adjustment Exploratory Protocols and Functional Evaluation of New Non Invasive Devices in Patient Volunteers
Acronym: MAP-EFNI PV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MAP-EFNI PV
Record Dates: First submitted 2016-05-12; First posted 2016-06-03 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Neurological Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (Experimental): Imaging devices
  Interventions: Device: Imaging devices

INTERVENTIONS:
Device: Imaging devices — technological adjustment tests

SUMMARY:
Parameters, sequences or paradigms optimisation in view of data quality and relevancy improvement.

DETAILED DESCRIPTION:
Various tests are needed for methodological optimization of the several devices (per-operative MRI, MEG, EEG, SPECT-CT, motor platform) of the technological platform.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers patient
* Male or female aged over 18 years
* Registered in the French social security scheme
* Signed informed consent

Exclusion Criteria:

* Contraindication to Magnetoencephalography (MEG) and/or Electroencephalography (EEG)
* Contraindication to Magnetic resonance imaging (MRI)
* All categories of protected persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-10-22 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Magnetic brain activity | 2 hours
  MEG records
Brain imaging | 2 hours
  MRI and SPECT-CT records
Electrical brain activity | 2 hours
  EEG records
Motor activity parameters | 2 hours
  Motor platform records

CONTACTS AND LOCATIONS:
Locations (1):
- CLINATEC, Grenoble, France

IPD SHARING:
Plan to Share IPD: No